CLINICAL TRIAL: NCT03140319
Title: Autologous Transplantation of Cultured Fibroblast for Correction of Nasolabial Folds
Brief Title: Transplantation of Fibroblast for Correction of Nasolabial Folds
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SCARM Institute, Tabriz, Iran (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCARM-Skin-001
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-07

CONDITIONS: Nasolabial Folds; Skin Aging
Keywords: Fibroblast; Cell transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibroblast (Experimental): Injection of Fibroblast
  Interventions: Biological: Fibroblast
- Placebo (Placebo Comparator): the patient receive placebo injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fibroblast — Transplantation of 20 million cell by three injection
  Other Names: Autologous injection of Fibroblast
  Arms: Fibroblast
Biological: Placebo — Injection of Placebo
  Arms: Placebo

SUMMARY:
The study evaluated the safety and efficacy of the Autologous cultured fibroblast for correction of Nasolabial folds and inhibition of skin aging

DETAILED DESCRIPTION:
Autologous cultured fibroblast which is obtain from the patient's normal skin is harvested and expanded in an in vitro. Biopsies samples are obtained from the behind of the patient's ear as a source of fibroblasts, then fibroblast cells isolated and expanded through cell culture, and used for the correction of Nasolabial folds, deep wrinkles of the forehead. Prior to final packaging, cell viability is assessed to be at least 85%

ELIGIBILITY:
Inclusion Criteria:

* Available and willing to attend all follow-up visits.
* Age > 18 years.
* Able and willing to give informed consent

Exclusion Criteria:

* Known allergy or sensitivity to any cellular products
* The subject has received a soft tissue augmentation to the area to be treated within the last 6 months.
* Subject is unwilling to forgo any cosmetic augmentation procedures for the duration of the study.
* The subject has received autologous fat transfer in the last 6 months.
* Subject is suffering from facial Kaposi's sarcoma.
* The subject has active skin diseases or inflammation on or near the area of injection
* positive HIV, hepatitis B virus (HBV), hepatitis C virus (HCV)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-10 (Estimated); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-26 (Estimated)

PRIMARY OUTCOMES:
Correction of Nasolabial | 6 months after transplantation
  Evaluate the correction of skin changes after transplantation of autologous fibroblasts by medical examination

CONTACTS AND LOCATIONS:
Overall Officials: Peyman Keyhanvar, MD, Ph.D, Study Director — Deputy for translational medicine of SCARM institute; Mohammad Nouri, Ph.D, Study Chair — Head of SCARM institute; Raheleh Farahzadi, Ph.D, Principal Investigator — cardiovascular research center, Tabriz University of Medical Sciences, Tabriz, Iran; Samira Asghari, MSc, Principal Investigator — SCARM institute
Locations (1):
- Stem cell and Regenerative Medicine institute (SCARM), Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss RA, Weiss MA, Beasley KL, Munavalli G. Autologous cultured fibroblast injection for facial contour deformities: a prospective, placebo-controlled, Phase III clinical trial. Dermatol Surg. 2007 Mar;33(3):263-8. doi: 10.1111/j.1524-4725.2007.33060.x. PMID 17338681
- [Result] Munavalli GS, Smith S, Maslowski JM, Weiss RA. Successful treatment of depressed, distensible acne scars using autologous fibroblasts: a multi-site, prospective, double blind, placebo-controlled clinical trial. Dermatol Surg. 2013 Aug;39(8):1226-36. doi: 10.1111/dsu.12204. Epub 2013 Apr 8. PMID 23566237
- [Result] Purdue GF, Hunt JL, Still JM Jr, Law EJ, Herndon DN, Goldfarb IW, Schiller WR, Hansbrough JF, Hickerson WL, Himel HN, Kealey GP, Twomey J, Missavage AE, Solem LD, Davis M, Totoritis M, Gentzkow GD. A multicenter clinical trial of a biosynthetic skin replacement, Dermagraft-TC, compared with cryopreserved human cadaver skin for temporary coverage of excised burn wounds. J Burn Care Rehabil. 1997 Jan-Feb;18(1 Pt 1):52-7. doi: 10.1097/00004630-199701000-00009. PMID 9063788
- [Result] Rigotti G, Charles-de-Sa L, Gontijo-de-Amorim NF, Takiya CM, Amable PR, Borojevic R, Benati D, Bernardi P, Sbarbati A. Expanded Stem Cells, Stromal-Vascular Fraction, and Platelet-Rich Plasma Enriched Fat: Comparing Results of Different Facial Rejuvenation Approaches in a Clinical Trial. Aesthet Surg J. 2016 Mar;36(3):261-70. doi: 10.1093/asj/sjv231. PMID 26879294